CLINICAL TRIAL: NCT02548845
Title: An Observational, Retrospective Study to Describe the Extent of Adherence to the Spanish Society of Medical Oncology Algorithm for the Treatment of Hyponatraemia Secondary to SIADH in Oncology Patients in Spain (ALGA)
Brief Title: An Observational Study to Describe the Adherence to the SEOM Algorithm for the Treatment of Hyponatraemia in Spain
Acronym: ALGA
Status: Completed | Type: Observational
Sponsor: Otsuka Pharmaceutical Europe Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 156-303-00043
Record Dates: First submitted 2015-09-07; First posted 2015-09-14 (Estimated); Results first posted 2018-08-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2017-11

CONDITIONS: Hyponatremia; Syndrome of Inappropriate ADH (SIADH) Secretion
Keywords: hyponatremia; SIADH; Oncologic patients
MeSH Terms: conditions — Hyponatremia; Inappropriate ADH Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In 2014, the Spanish Sociedad Española de Oncología Médica (SEOM) algorithm for the treatment of hyponatraemia secondary to to syndrome of inappropriate antidiuretic hormone (SIADH) in oncology patients was developed. Since it is hypothesised that the adherence to the SEOM algorithm is not 100%, the current retrospective non-interventional study will investigate the perceived and actual adherence of participating centres to the SEOM algorithm and its impact on patient outcomes

ELIGIBILITY:
Inclusion Criteria:

* Provision of patient informed consent unless a) not required by local regulations, b) it would represent a non-reasonable effort or c) if the source patient is deceased or untraceable.
* Female and/or male oncology patients aged 18 years and over
* Patients who have experienced at least one occurrence of hyponatraemia secondary to the SIADH.

Exclusion Criteria:

* A patient cannot take part in this study if participating in any clinical study in which the medicinal product aims to treat the causes or symptoms of hyponatraemia at the time of the hyponatraemia episode being documented in the current study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients are oncology patients ≥ 18 years old who had been diagnosed with at least one occurrence of hyponatraemia secondary to the SIADH and who had been managed ein one of the Spanish centres who have implemented the SEOM algorithm.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2015-12; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Department, Study Director — Otsuka Europe
Locations (4):
- Spain (4):
  - Castellon
  - Madrid
  - Santiago de Compostela
  - Seville

RESULTS

PARTICIPANT FLOW:
Groups:
- Oncology Patients With Hyponatraemia: Adult oncology patients who have been treated for ≥ 1 episode of hyponatraemia secondary to the SIADH (defined as a serum sodium level <135 mmol/L)
Period: Overall Study
Arm/Group | Oncology Patients With Hyponatraemia
Started | 70
Completed | 70
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Oncology Patients With Hyponatraemia
Number analyzed (Participants) | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (13.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 49
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 70
Weight [Mean (Standard Deviation); unit: kg] | 68.4 (13.00)
Height [Mean (Standard Deviation); unit: meters] | 1.656 (0.1031)
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 25.075 (4.3126)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Managed According to the SEOM Algorithm (as a Result Adherence to the Algorithm Will be the % of These Patients Among the Total Number of Patients)
Description: Adherence to the algorithm will be evaluated using a pre-defined decision tree that will be provided in the electronic case report form (eCRF) and will be completed by the investigator
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 4 days (follow-up will stop after a maximum of 6 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Oncology Patients With Hyponatraemia
Number analyzed (Participants) | 70
Participants | 20

2. Secondary Outcome: Time to Sodium Level Improvement for Patients Who Were and Were Not Treated in Adherence With the SEOM Algorithm (Days)
Description: Improvement is defined as a change in the baseline sodium level category (mild, moderate or severe) from a worse category to a better category or eunatraemia. Note that the time to improvement of sodium levels was defined as the first date/time of improvement of sodium levels - date/time of collection of serum sodium levels at baseline (for patients where there was an improvement in sodium levels) or as the final date/time of collection of serum sodium levels - date/time of collection of serum sodium levels at baseline (for patients that did not achieve an improvement in sodium levels [censored patients]).
Time Frame: Longitudinal (up to discharge or a maximum of 6 weeks after onset of hyponatremia episode)
Population: The overall number of patients analysed represents the number of participants for which the data (time in days) was available. As a retrospective chart review, there were some missing data in this outcome measure (date of improvement in this case)
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Participants Treated According to SEOM Algorithm: Adult oncology patients who have been treated for ≥ 1 episode of hyponatraemia secondary to the SIADH according to the SEOM algorithm.
- Participant NOT Treated According to SEOM Algorithm: Adult oncology patients who have been treated for ≥ 1 episode of hyponatraemia secondary to the SIADH not according to the SEOM algorithm.
Arm/Group | Participants Treated According to SEOM Algorithm | Participant NOT Treated According to SEOM Algorithm
Number analyzed (Participants) | 19 | 47
Days | 5 [3 to 15] | 4 [2 to 7]

3. Secondary Outcome: Time to Initiation or Re-initiation of Chemotherapy (Since the Start of the Hyponatraemia Episode) in Patients Candidate for Chemotherapy Who Were and Were Not Treated in Adherence With the SEOM Algorithm.
Time Frame: Longitudinal (up to discharge or a maximum of 6 weeks after onset of hyponatremia episode)
Population: In this analysis, only the 22 patients who were candidate for chemotherapy during the study period were included, this explains the difference with the total number of participants.
Measure: Median (95% Confidence Interval); unit: Hours
Groups:
- Subjects With Chemotherapy Treated as Per SEOM Algorithm: Adult oncology patients who have been treated for ≥ 1 episode of hyponatraemia secondary to the SIADH according to the SEOM algorithm and who were candidate for or actually in chemotherapy treatement when the hyponatremia episode occurred.
- Subjects With Chemotherapy NOT Treated as Per SEOM Algorithm: Adult oncology patients who have been treated for ≥ 1 episode of hyponatraemia secondary to the SIADH NOT according to the SEOM algorithm and who were candidate for or actually in chemotherapy treatement when the hyponatremia episode occurred
Arm/Group | Subjects With Chemotherapy Treated as Per SEOM Algorithm | Subjects With Chemotherapy NOT Treated as Per SEOM Algorithm
Number analyzed (Participants) | 8 | 14
Hours | 14.5 [5 to 35] | 15.5 [7 to 181]

4. Secondary Outcome: Length of Hospitalisation (Measured From the Start of the Hyponatraemia Episode to Discharge) for Patients Who Were and Were Not Treated in Adherence With the Algorithm
Time Frame: Longitudinal (up to discharge or a maximum of 6 weeks after onset of hyponatremia episode)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Participants Treated According to SEOM Algorithm | Participant NOT Treated According to SEOM Algorithm
Number analyzed (Participants) | 20 | 50
Days | 16.5 [8 to 27] | 9.5 [7 to 22]

5. Secondary Outcome: Time to Sodium Level Improvement for Patients Who Were and Were Not Treated in Adherence With the SEOM Algorithm (Hours)
Description: as for outcome 2
Time Frame: Longitudinal (up to discharge or a maximum of 6 weeks after onset of hyponatremia episode)
Population: The overall number of patients analysed represents the number of participants for which the data (time in hours) was available. As a retrospective chart review, there were some missing data in this outcome measure (time of improvement in this case)
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Participants Treated According to SEOM Algorithm | Participant NOT Treated According to SEOM Algorithm
Number analyzed (Participants) | 17 | 15
hours | 80.5 [38.3 to 331.4] | 134.6 [33.2 to 444.9]

ADVERSE EVENTS:
Time Frame: From the onset of the hyponatraemia episode until 6 weeks afterwards
Description: Any untoward medicinal occurrence in a patient administered a medicinal product and which does not necessarily have a causal relationship with this treatment (Directive 2001/83/EC amended by Directive 2010/ 84/ EU). An AE can therefore be any unfavourable and unintended sign (e.g., abnormal laboratory finding), symptom or disease temporally associated with the use of a medicinal product, whether or not it is considered causally related to the medicinal product.
Arm/Group | Oncology Patients With Hyponatraemia
All-Cause Mortality (participants affected / at risk) | 5/70
Serious Adverse Events (participants affected / at risk) | 10/70
Other Adverse Events (participants affected / at risk) | 7/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oncology Patients With Hyponatraemia (N=70)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (1)
Listless (Psychiatric disorders) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Death (General disorders) | 2 (2)
Delirium (Psychiatric disorders) | 1 (1)
General physical health deterioriation (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oncology Patients With Hyponatraemia (N=70)
Constipation (Gastrointestinal disorders) | 2 (2)
Pain (General disorders) | 2 (2)
Asthenia (General disorders) | 2 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Recruitment problems leading to smaller sample size than expected (70 patients vs 100). A priori, the impact on precision was considered acceptable (95% confidence interval equal to ± 10.0% with 100 patients vs ± 11.7% with 70 patients).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
As a multicentre study, the first publication shall be based on consolidated analysed data from all centres, i.e. the publication of results from individual institution/Investigator is not allowed before the publication of the full study results.

The PI agrees to give the sponsor 60 days to review the communications. If case of propietary information inadvertenly divulged, intellectual property rights at risk or inaccurate information presented, changes can be required by the sponsor.